CLINICAL TRIAL: NCT04443894
Title: Acute & Chronic Post-mastectomy Pain: Can PECS Block Alter the Geography?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Chrysanthi Batistaki, Associate Professor of Anaesthesiology, Attikon Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BreastPecs
Record Dates: First submitted 2020-06-21; First posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Immediate and Chronic Pain After Mastectomy Managed With PECS Block or Local Infiltration
Keywords: pain; mastectomy; PECS
MeSH Terms: conditions — Pain | interventions — Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: PATIENT OUTCOME ASSESSOR
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PECS block (Active Comparator)
  Interventions: Other: PECS block
- local infiltration (Active Comparator)
  Interventions: Other: local infiltration

INTERVENTIONS:
Other: PECS block — PECS block is performed at the side of surgery (II) before incision with ropivacaine 0,375%.(30 ml). General anesthesia is induced and maintained with midazolam, fentanyl, propofol and rocuronium. Pain is assessed postoperatively according to protocol (24 hours and after 3 months).
  Arms: PECS block
Other: local infiltration — local infiltration of the surgical wound before incision with πwith ropivacaine 0,375%.(30 ml). General anesthesia is induced and maintained with midazolam, fentanyl, propofol and rocuronium. Pain is assessed postoperatively according to protocol (24 hours and after 3 months).
  Arms: local infiltration

SUMMARY:
Post mastectomy pain management is of crucial importance for patients' rehabilitation and quality of life. PECS block is used for acute and chronic post mastectomy pain management. Surgical infiltration is also used in this field. Patients in our study are divided in two groups receiving PECS block or surgical infiltrationbefore incision. Multimodal analgesia is indispensable according to recent guidelines for enhanced postoperative recovery. Pain scores will be assessed during the first 24h postoperatively and at 3 months after surgery.

DETAILED DESCRIPTION:
Patients are randomly assigned to 2 groups, PECS block or surgical infiltration group. Patients assigned to PECS group will receive 30cc of ropivacaine 0,375% where 10cc will be injected between pectoralis major and pectoralis minor and 20cc between pectoralis minor and serratus anterior muscle under ultrasound guidance. Patients assigned to surgical infiltration group will receive 30cc of ropivacaine 0,375% injected by the surgeon. Local aneshetic is administered in both groups after the induction of general anesthesia and before incision. Pain will be assessed at 1, 12, 24h after surgery and at three months after surgery communicating by telephone. Post operative analgesia includes paracetamol 1gr, parecoxib 40 mg (as required) and tramadol as rescue analgesia (1 mg/kg iv up to 3 times daily). Chronic pain will be assessed after 3 months as for prevalence and neuropathic characteristics.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* ASA physical status I-III
* elective partial mastectomy

Exclusion Criteria:

* refusal of patient participation or inability to participate to the study

  * known allergic reaction to drugs included in the study design
  * contraindiations of performance of peripheral regional anesthesia
  * diabetes melitus or known neurological disorder
  * chronic pain disorders under therapy with opioids or other analgesic drugs for chronic pain
  * all male patients
  * all patients not speaking the Greek language

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — only women
Enrollment: 40 (Estimated)
Dates: Start 2020-05-20 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
intensity of acute postoperative pain | 24 hours
  intensity of acute postoperative pain, numeric rating scale 0-10

SECONDARY OUTCOMES:
intensity of chronic pain | 3 months
  intensity of chronic pain with numeric rating scale 0-10
Prevalence of chronic neuropathic pain | 3 months
  Prevalence of chronic pain at the site of surgery, measured with the LANSS questionnaire
Prevalence of chronic neuropathic pain | 3 months
  Prevalence of chronic pain at the site of surgery, measured with YES./NO

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Department of Anesthesiology, Attikon Hospital, 1 Rimini str., Athens, Greece

IPD SHARING:
Plan to Share IPD: No